CLINICAL TRIAL: NCT06530862
Title: Comparison of the Efficacy of ESWT and Dry Needling Treatments in the Management of Piriformis Syndrome; A Randomized Study
Brief Title: Piriformis Syndrome; Extracorporeal Shock Wave Therapy and Dry Needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Burak Tayyip Dede, Medical Doctor, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22/12/2023; 2011-KAEK-50;347
Record Dates: First submitted 2024-07-27; First posted 2024-07-31 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Piriformis Syndrome; Extracorporeal Shock Wave Therapy
Keywords: ESWT; Dry Needling; Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into 2 groups and will be treated with ESWT or Dry needling
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT group (Active Comparator): Patients in this group received three sessions of ESWT at an energy density of 4 bars and a frequency of 2,000 shocks/min at 5 Hz for three weeks, each session once a week.
  Interventions: Other: ESWT+stretching exercises
- Dry needling (Active Comparator): The piriformis muscle of the patients in the group will be dry needled with 0.6*80 mm acupuncture needles under ultrasound guidance for 3 sessions at one week intervals.
  Interventions: Other: Dry needling+stretching exercises

INTERVENTIONS:
Other: ESWT+stretching exercises — Participants in this group will receive ESWT treatment
  Arms: ESWT group
Other: Dry needling+stretching exercises — Participants in this group will receive Dry needling treatment
  Arms: Dry needling

SUMMARY:
This study is being conducted on patients with piriformis syndrome. Patients are divided into two groups by list randomization method: Extracorporeal shock wave therapy (ESWT) group and Dry neddling (DN) group. Both groups of patients agreed to perform basic stretching exercises. The ESWT group received 3 sessions of radial ESWT, 1 session per week. The DN group received 3 sessions of ultrasound-guided needling, 1 session per week. Clinical evaluations of the participants were performed at the beginning of treatment, 1 month, and 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Complaint for more than 3 months

Exclusion Criteria:

* disc pathologies according to radiological imaging
* hip joint and soft tissue pathologies
* recent history of trauma, history of surgery in the lumbar and hip region
* history of rheumatologic disease
* history of polyneuropathy
* history of sciatic nerve injury
* history of malignancy
* opioid analgesia or corticosteroid intervention for pain in the last month
* patients receive another treatment during the study
* Having a contraindication for DN treatment or ESWT treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-02-03 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) score | 7 months
  Pain was evaluated with a Visual analog scale (VAS) score
Lower extremity functiunal scale (LEFS) | 7 months
  Pain was evaluated with a Lower extremity functiunal scale (LEFS (minimum=0, maximum=80)) The higher the score, the better the result
Oswestry disability index (ODI) | 7 months
  Pain was evaluated with a Oswestry disability index (ODI (minimum=0, maximum=60))The lower the score the better the result

CONTACTS AND LOCATIONS:
Locations (1):
- Burak Tayyip Dede, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No